CLINICAL TRIAL: NCT06663917
Title: Clinical Evaluation of Frequency Allocation for Bimodal CI Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-00833; R01DC021980-01 (NIH)
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experienced Users (Experimental): All subjects will be fit with a modified cochlear implant program ("experimental FAT") that changes which frequencies are presented to the cochlear implant. Subjects will complete a 1 month adaptation to the experimental FAT (438 Hz) and then a one month re-adaptation to the standard FAT (188 Hz). Speech perception tests and questionnaires will be collected before and after each FAT adaptation.
  Interventions: Other: Experimental frequency allocation table (FAT) - 438 Hz; Other: Standard FAT - 188 Hz

INTERVENTIONS:
Other: Experimental frequency allocation table (FAT) - 438 Hz — The modified cochlear implant program ("experimental FAT") changes which frequencies are presented to the cochlear implant. The experimental FAT frequency of 438 Hz will be loaded onto the subjects processor via the CI Select Mobile App. Subjects will use the experimental FAT for one month.
Other: Standard FAT - 188 Hz — All subjects will retain one program with the standard 188 Hz FAT. Subjects will use the standard FAT for one month.

SUMMARY:
This study will examine experienced, bimodal cochlear implant (CI) patients who receive an alternative frequency allocation table (FAT) to determine how it improves sound quality, device satisfaction, and speech perception abilities with respect to the standard default FAT. The goal of this study is to investigate how improving place-pitch mismatch in bimodal CI users affects 1) sound quality, 2) satisfaction, and 3) speech perception.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Regular usage of a cochlear implant device with at least 18 active electrodes, and compliance with programming/appointments
3. Received a cochlear implant at least 6 months ago and use a hearing aid in the contralateral ear
4. Pure tone average (.5, 1, and 2kHz) between 30 and 70 dB (decibel) hearing level in the contralateral (hearing aid) ear
5. Standard FAT use for all programs prior to study participation
6. No known anatomical abnormalities in either ear
7. English speaking
8. No known cognitive impairments
9. At least 25% of subjects should use the Cochlear EA32 electrode

Exclusion Criteria:

1. Under age 18
2. Non-English speaking. Participants that are Non-English speaking are excluded from this study due to the use of speech testing materials that are validated in the English language. Additionally, study team members are not equipped to appropriately score speech testing materials validated in other languages.
3. Cognitively impaired
4. Non-consistent device usage
5. Greater than 70 dB hearing level pure tone average in the contralateral ear
6. Normal hearing or mild hearing loss in the contralateral ear
7. Non-standard FAT programs
8. Use of any frequency transposition programming in hearing aid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-06 (Actual); Primary Completion 2027-10-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
Sound Quality Questionnaire Score while using standard 188 Hz FAT | Baseline
  A questionnaire will be given to the subjects to record their subjective thoughts regarding sound quality and satisfaction with both the experiment FAT and the standard FAT. Questionnaires will be administered double blind. Patients evaluate the 16-item questionnaire using a likert-scale (1-strongly disagree to 5-strongly agree). Lower scores indicate decreased sound quality and satisfaction, while higher scores indicate increased sound quality and satisfaction.
Sound Quality Questionnaire Score while using experimental 438 Hz FAT | Behavioral Visit 2 (1 month post 438 Hz FAT adaptation)
  A questionnaire will be given to the subjects to record their subjective thoughts regarding sound quality and satisfaction with both the experiment FAT and the standard FAT. Questionnaires will be administered double blind. Patients evaluate the 16-item questionnaire using a likert-scale (1-strongly disagree to 5-strongly agree). Lower scores indicate decreased sound quality and satisfaction, while higher scores indicate increased sound quality and satisfaction.
Sound Quality Questionnaire Score while using standard 188 Hz FAT | Behavioral Visit 3 (1 month post 188 Hz FAT re-adaptation)
  A questionnaire will be given to the subjects to record their subjective thoughts regarding sound quality and satisfaction with both the experiment FAT and the standard FAT. Questionnaires will be administered double blind. Patients evaluate the 16-item questionnaire using a likert-scale (1-strongly disagree to 5-strongly agree). Lower scores indicate decreased sound quality and satisfaction, while higher scores indicate increased sound quality and satisfaction.
The consonant-nucleus-consonant (CNC) word list score while using standard 188 Hz FAT | Baseline
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CNC word list score while using standard 188 Hz FAT | Behavioral Visit 2 (1 month post 438 Hz FAT adaptation)
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CNC word list score while using standard 188 Hz FAT | Behavioral Visit 3 (1 month post 188 Hz FAT re-adaptation)
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CNC word list score while using experimental 438 Hz FAT | Baseline
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CNC word list score while using experimental 438 Hz FAT | Behavioral Visit 2 (1 month post 438 Hz FAT adaptation)
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CNC word list score while using experimental 438 Hz FAT | Behavioral Visit 3 (1 month post 188 Hz FAT re-adaptation)
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score using standard 188 Hz FAT | Baseline
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score using standard 188 Hz FAT | Behavioral Visit 2 (1 month post 438 Hz FAT adaptation)
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score using standard 188 Hz FAT | Behavioral Visit 3 (1 month post 188 Hz FAT re-adaptation)
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score using experimental 438 Hz FAT | Baseline
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score using experimental 438 Hz FAT | Behavioral Visit 2 (1 month post 438 Hz FAT adaptation)
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score using experimental 438 Hz FAT | Behavioral Visit 3 (1 month post 188 Hz FAT re-adaptation)
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A. Svirsky, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Data are available indefinitely in Databrary database (Link to be included when database is created). The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Data are available indefinitely in Databrary database (Link to be included when database is created). To gain access, data requestors will need to sign a data access agreement.